CLINICAL TRIAL: NCT05114330
Title: Non-interventional, Prospective Observational Study of the Treatment Practice of CNS Involvement of Malignant Lymphoma in Routine Clinical Practice
Brief Title: Secondary Central Nervous System Lymphoma Registry - Charité
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Stefan Habringer, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: SZNSL-R
Record Dates: First submitted 2021-10-25; First posted 2021-11-09 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Central Nervous System Lymphoma; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood, tumor tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Systemic (= localized outside the CNS) lymphoma with secondary CNS involvement at initial diagnosis
- Cohort 2: CNS relapse of previously systemic lymphoma

SUMMARY:
The objective of the observation is to collect and document data on treatment strategies for secondary central nervous system lymphoma (SCNSL) in routine clinical practice, whether obtained in the context of clinical trials or outside of trials. In particular, the following questions will be specified:

* What therapeutic approaches are being pursued?
* What is the clinical outcome of the various treatment options?
* What is the frequency of serious adverse events with each therapeutic approach?

DETAILED DESCRIPTION:
The observational study is to be conducted in inpatient clinics, outpatient clinics and by oncology physicians in private practice. The investigators will be invited to participate by the Charité - CNS Lymphoma Working Group (Charité AG ZNSL) or the Competence Network Malignant Lymphomas (KML). When a patient is reported, the personal data of the physician including the patient will be recorded and compiled in the form of a list documentation.

All patients with SCNSL can and should be included in the study regardless of which therapy options are used and regardless of whether it is a first-line treatment, the treatment of a recurrence or a maintenance therapy for SCNSL. No intervention is associated with the conduct of the observational study with regard to the selection and implementation of the specific therapeutic regimen, diagnostics, and examination frequency during and after treatment.

The following information should be documented:

* Patient demographics and medical history
* Tumor extent at the time of initial diagnosis and CNS involvement
* Prior therapy
* General condition
* Therapy regimen for the CNS involvement
* Response
* Adverse drug reactions
* Tolerability of therapy: acute toxicity
* Chronic therapy toxicity, especially late neurotoxicity
* Time to treatment failure (relapse or progression)
* Death from any cause

ELIGIBILITY:
Inclusion Criteria:

• All patients with SCNSL can and should be included in the registry regardless of which treatment options are used and whether the treatment being given is first-line, recurrence, or maintenance therapy for SCNSL.

Exclusion Criteria:

• None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with SCNSL
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-06-08 (Actual); Primary Completion 2024-06-08 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
Description of different therapeutic regimens | Through study completion, an average of 3 years
  Description of different therapeutic regimens
Outcome of different therapeutic regimens | Through study completion, an average of 3 years
  Overall Survival
Outcome of different therapeutic regimens | Through study completion, an average of 3 years
  Progression Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin, Med. Klinik m. S. Hämatologie, Onkologie und Tumorimmunologie (CBF), Berlin, Germany

REFERENCES:
- [Derived] Habringer S, Demel UM, Fietz AK, Lammer F, Schroers R, Hofer S, Bairey O, Braess J, Meier-Stiegen AS, Stuhlmann R, Schmidt-Hieber M, Hoffmann J, Zinngrebe B, Kaiser U, Reimer P, Mohle R, Fix P, Hoffkes HG, Langenkamp U, Buschenfelde CMZ, Hopfer O, Stoltefuss A, La Rosee P, Blasberg H, Jordan K, Kaun S, Meurer A, Unteroberdorster M, von Brunneck AC, Capper D, Heppner FL, Chapuy B, Janz M, Schwartz S, Konietschke F, Vajkoczy P, Korfel A, Keller U. A prospective observational study of real-world treatment and outcome in secondary CNS lymphoma. Eur J Cancer. 2024 Jan;196:113436. doi: 10.1016/j.ejca.2023.113436. Epub 2023 Nov 14. PMID 38008033